CLINICAL TRIAL: NCT06182254
Title: Personalized Perioperative Care Based on Patient Reported Outcomes Measures: Randomized Controlled Trial Based on the QoR-15
Brief Title: Personalized Perioperative Care Based on Patient Reported Outcomes Measures
Acronym: SUPPORT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 8801
Record Dates: First submitted 2023-04-06; First posted 2023-12-26 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Surgery; Perioperative Medicine
Keywords: perioperative; surgery; care Patient Reported Outcomes Measures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group: OPTIMISTIC follow-up (Experimental): follow-up by nurses specialized in collecting the patient's point of view concerning his or her state of health, in addition to the usual conventional follow-up according to routine care directive interviews carried out preoperatively and at Days 1, 3, 14 and 28 postoperatively (modified QoR-15f score, PROMS...)
  Interventions: Behavioral: Experimental group: OPTIMISTIC follow-up
- Control group: Usual conventional follow-up (Active Comparator): usual conventional follow-up according to routine care (modified QoR-15f score will be administered to all patients at visit 0 and Day 35).
  Interventions: Other: Control group: Usual conventional follow-up

INTERVENTIONS:
Behavioral: Experimental group: OPTIMISTIC follow-up — follow-up by nurses specialized in collecting the patient's point of view concerning his or her state of health, in addition to the usual conventional follow-up according to routine care directive interviews carried out preoperatively and at Days 1, 3, 14 and 28 postoperatively (modified QoR-15f score, PROMS...)
  Arms: Experimental group: OPTIMISTIC follow-up
Other: Control group: Usual conventional follow-up — usual conventional follow-up according to routine care (modified QoR-15f score will be administered to all patients at visit 0 and Day 35).
  Arms: Control group: Usual conventional follow-up

SUMMARY:
In the perioperative setting, Patient Reported Outcomes Measures (PROMs) are important for both patients and clinicians.

Reliable PROMs, like the Quality Of Recovery 15 (QoR-15) questionnaire, are available for patients experiencing surgery. These PROMs are significantly used as endoints for clinical interventions assessment. These PROMs may also be considered to monitor and assess patient health status as part of enhanced recovery after surgery pathway.

However data about the efficacy of PROMs-based perioperative clinical follow up are lacking.

The clinical hypothesis is that a PROMs (QoR-15) based perioperative clinical care is more efficient that the usual care non based on the QoR-15.

DETAILED DESCRIPTION:
The study is a multicenter randomized controlled trial comparing 2 groups:

* A control group, including the usual conventional follow-up by the surgeon and the attending physician.
* An experimental group including, in addition to the usual conventional follow-up, the follow-up by nurses specialized in the evaluation of the PROMs using the french version of the QoR-15 questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* adult patient
* Benefiting from an osteo-articular surgery
* Subject affiliated to a social health insurance plan
* Able to understand the objectives and risks of the research and to give a dated and signed informed consent

Exclusion Criteria:

* Inability to administer the QoR-15f questionnaire (cognitive impairment, language barrier)
* Subject under court protection
* Subject under guardianship or curatorship
* Patient whose rehabilitation will be performed in a secondary hospital
* Patient having already benefited from a previous follow-up by the OPTIMISTE team
* Patient included in a therapeutic trial that may impact postoperative quality of recovery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2023-04-14 (Actual); Primary Completion 2025-01-23 (Actual); Study Completion 2025-01-23 (Actual)

PRIMARY OUTCOMES:
Evaluate the effectiveness of a perioperative follow-up integrating the patient's point of view in osteoarticular surgery compared to a classic postoperative management | Inclusion (Day 0), Day 1, Day 3, Day 14, Day 28 and Day 35
  Evolution of a modified version of the French Quality-Of-Recovery 15 score (QoR-15f) between the intraoperative consultation and D35 postoperative

SECONDARY OUTCOMES:
Describe postoperative functional recovery after osteoarticular surgery | Inclusion (Day 0), Day 1, Day 3, Day 14, Day 28 and Day 35
  Isolated and dimensional changes in the 15 items of the QoR-15f score from intraoperative consultation to postoperative D35.
Describe the consequences of a perioperative follow-up that integrates the patient's point of view on the patient pathway | Day 1, Day 3, Day 14, Day 28 and Day 35
  Number of medical and paramedical consultations and number of hospitalization days between hospital discharge and D35 postoperative
Evaluate the effectiveness of perioperative monitoring that incorporates the patient's perspective on reducing postoperative opioid use | Day 35
  Opioid consommation at D35 postoperative
Evaluate the safety | Inclusion (Day 0), Day 1, Day 3, Day 14, Day 28 and Day 35]
  postoperative complication rate to postoperative D35

CONTACTS AND LOCATIONS:
Overall Officials: EBER Manon, Mme, Principal Investigator — CHRU Strasbourg
Locations (1):
- EBER Manon, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No